CLINICAL TRIAL: NCT04473157
Title: Detection of SARS-CoV-2 in Patients Presenting With Anosmia During COVID-19 Pandemic Era in Egypt
Brief Title: COVID-19 in Patients With Anosmia in Egypt
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ossama Mansour, MD, FACS, Professor of Otolaryngology, Ain Shams University
Other Study IDs: FMASU P45a/2020
Record Dates: First submitted 2020-07-15; First posted 2020-07-16 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Anosmia; Covid19; Dysgeusia
Keywords: Corona virus; SARS-CoV-2; Olfactory Disturbance; Taste Disturbance
MeSH Terms: conditions — Anosmia; COVID-19; Dysgeusia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasopharyngeal and oropharyngeal Swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to test the frequency of severe acute respiratory syndrome new corona virus SARS-CoV-2 or other respiratory viruses in patients presenting with anosmia or dysgeusia to Ain Shams University Hospitals, Cairo, Egypt.

DETAILED DESCRIPTION:
Fifty Patients presenting to Triage and/or Ear, Nose and Throat (ENT) clinics in Ain Shams University Hospitals with the chief complaint of Anosmia/ dysgeusia in the period July- September 2020; will undergo thorough history taking, clinical assessment and polymers chain reaction rt-PCR to SARS-COV2; and if proven negative to COVID 19, PCR to other respiratory pathogens will be tested. COVID-19 patients will be managed according to the standard protocol of Ain Shams University Hospitals. Follow up after 3 weeks for the outcome of recovery of the smell sense and seroconversion by rapid test for immunoglobulins IgM/ IgG of COVID 19, for the probability of a false negative PCR at initial visit.

Ethical committee approval for the current study protocol was obtained. Patients will be invited to participate and the informed consent will be signed.

ELIGIBILITY:
Inclusion Criteria:

* adult (>18 years) patients presented with acute-onset anosmia.

Exclusion Criteria:

* patients with anosmia or gustatory dysfunctions before the epidemic; patients with previous history of chronic sinusitis or previous sinus surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fifty Patients presenting to Triage and/or ENT clinics in Ain Shams University Hospitals with the chief complaint of Anosmia/ dysgeusia in the period July- August 2020
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Recovery from Anosmia | 3 weeks
  subjective questionnaire about smell and taste
Seroconversion | 3 weeks
  developing IgM/ IgG antibodies by rapid test

SECONDARY OUTCOMES:
COVID 19 | 3 weeks
  developing other symptoms of COVID 19

CONTACTS AND LOCATIONS:
Overall Officials: Ossama I Mansour, MD, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

REFERENCES:
- [Background] Moein ST, Hashemian SM, Mansourafshar B, Khorram-Tousi A, Tabarsi P, Doty RL. Smell dysfunction: a biomarker for COVID-19. Int Forum Allergy Rhinol. 2020 Aug;10(8):944-950. doi: 10.1002/alr.22587. Epub 2020 Jun 18. PMID 32301284
- [Background] Spinato G, Fabbris C, Polesel J, Cazzador D, Borsetto D, Hopkins C, Boscolo-Rizzo P. Alterations in Smell or Taste in Mildly Symptomatic Outpatients With SARS-CoV-2 Infection. JAMA. 2020 May 26;323(20):2089-2090. doi: 10.1001/jama.2020.6771. PMID 32320008
- [Background] Menni C, Valdes AM, Freidin MB, Sudre CH, Nguyen LH, Drew DA, Ganesh S, Varsavsky T, Cardoso MJ, El-Sayed Moustafa JS, Visconti A, Hysi P, Bowyer RCE, Mangino M, Falchi M, Wolf J, Ourselin S, Chan AT, Steves CJ, Spector TD. Real-time tracking of self-reported symptoms to predict potential COVID-19. Nat Med. 2020 Jul;26(7):1037-1040. doi: 10.1038/s41591-020-0916-2. Epub 2020 May 11. PMID 32393804
- [Background] Desforges M, Le Coupanec A, Brison E, Meessen-Pinard M, Talbot PJ. Neuroinvasive and neurotropic human respiratory coronaviruses: potential neurovirulent agents in humans. Adv Exp Med Biol. 2014;807:75-96. doi: 10.1007/978-81-322-1777-0_6. PMID 24619619